CLINICAL TRIAL: NCT03375268
Title: Predictive Model for Postoperative Complications in Elderly Patients With Hip Arthroplasty: Retrospective Study
Brief Title: Predictive Model for Postoperative Complications in Hemi-hip Arthroplasty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-10-003
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Complication; Risk Factor; Elderly Patient; Arthroplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to identify the major complications and their risk factors of elderly patients who had undergone Hemi-hip Arthroplasty.

DETAILED DESCRIPTION:
We retrospectively reviewed the medical records and reviewed the major complications and identify risk factors of elderly patients who had undergone Hemi-hip Arthroplasty for adults aged 60 years or older from January 2011 to December 2015.

ELIGIBILITY:
Inclusion Criteria:

* A patient scheduled to undergo spinal anesthesia for Hemi-hip Arthroplasty

Exclusion Criteria:

* 1) Patients with acute infectious disease before surgery 2) Patients with fractures around the implant 3) Patients who underwent reoperation during hospitalization 4) During the study period, Duplicate patient who underwent the opposite side of the hip during hospitalization

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2011 to December 2015, we will enroll adult patients aged 60 years or older who underwent Hemi-hip Arthroplasty at our institution.
Sampling Method: Non-Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2011-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | from operation day to postoperative 30 days
  we collect postoperative complications which include cardiac, pulmonary renal, cerebral, and other complications.

CONTACTS AND LOCATIONS:
Overall Officials: Eunsu Choi, pf, Principal Investigator — Eulji University Hospital
Locations (1):
- Eulji university hospital, Seoul, South Korea